CLINICAL TRIAL: NCT03224065
Title: Randomized, Controlled Clinical Study of Non-tuberculosis Mycobacteria Lung Disease Treatment Based on GenSeizer Characteristic Gene Capture Strategy
Brief Title: NTM-LD Treatment Based on GenSeizer Characteristic Gene Capture Strategy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Haiqng Chu, Director, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K17-144
Record Dates: First submitted 2017-07-16; First posted 2017-07-21 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Non - Tuberculosis Mycobacteria Lung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recommended therapy group (No Intervention): Guideline recommended regimen for treatment, regardless of antibiotic resistant genotype test results
- Optimized therapy group (Experimental): Optimized therapy based on antibiotic resistant genotype test results
  Interventions: Diagnostic Test: Genotype detected through GenSeizer high-throughput gene capture technology

INTERVENTIONS:
Diagnostic Test: Genotype detected through GenSeizer high-throughput gene capture technology — The sputum and/or alveolar lavage fluid of the optimal treatment group was first identified by GenSeizer, which was used to remove the resistant agents and choose the sensitive agents, so as to optimize the initial antimicrobial program. All agents are within the recommended range of 2007 ATS / IDSA Guidelines. All treatment regimens need to be corrected in time according to the final results of culture and in vitro susceptibility testing.
  Arms: Optimized therapy group

SUMMARY:
Treatment of non - tuberculosis mycobacteria lung disease is challenging. The current treatment used is from 2007 American Thoracic Society guidelines recommended antibiotic combination therapy, which is lack of validation of clinical studies. More and more studies have confirmed that NTM antibiotic resistant gene will affect the efficacy, such as erm(41), rrl to clarithromycin, rrs to amikacin and so on. This study aimed to compare the efficacy of guideline recommended therapy and optimized therapy according to antibiotic susceptibility - related genotype.Genetic testing is accomplished through GenSeizer's high-throughput gene capture technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients met diagnostic criteria of NTM lung disease by ATS/IDSA on 2007
* non-CF Bronchiectasis

Exclusion Criteria:

* Already on treatment for NTM lung disease
* Appropriate exclusion of other lung diagnosis
* Patients with severe organ dysfunction

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Culture conversion rate | up to 18 months
  The proportion of final sputum conversion to culture negative

SECONDARY OUTCOMES:
Initial time of sputum culture conversion | up to 18 months
  The time of first sputum conversion to culture negative
Chest CT | up to 18 months
  Chest imaging changes of CT examination
Blood routine test | every month, up to 18months
liver function test | every month, up to 18months
kidney function test | every month, up to 18months

CONTACTS AND LOCATIONS:
Locations (1):
- Haiqing Chu, Shanghai, China